CLINICAL TRIAL: NCT04325659
Title: Evaluating a Neuromodulator Medical Device (Bridge Device) for Opioid Use Disorder Treatment
Brief Title: An Innovative Intervention for OUD Treatment
Acronym: Bridge
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00241133; R01DA048761 (NIH)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Opioid-Related Disorders; Opioid Dependence; Opioid Addiction; Opioid Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Intervention Model Description: The study is of a device (the Bridge Device), not of a drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Lofexidine/Sham Bridge Device (Active Comparator): Lofexidine (Lucemyra) encapsulated
  Interventions: Drug: Lofexidine; Device: Sham Bridge Device
- Sham Bridge Device /Placebo Study Drug (Placebo Comparator): Inactive Bridge Device and placebo study drug
  Interventions: Drug: Placebo; Device: Sham Bridge Device
- Active Bridge Device/ Placebo Study Drug (Experimental): Active Bridge Device and placebo study drug
  Interventions: Device: Bridge Device; Drug: Placebo

INTERVENTIONS:
Device: Bridge Device — An FDA-cleared neuromodulator medical device, marketed for the treatment of opioid withdrawal
  Other Names: NSS-2 Bridge Device
  Arms: Active Bridge Device/ Placebo Study Drug
Drug: Lofexidine — FDA-approved medication for the treatment of opioid withdrawal. Participants will receive capsules 4 times daily for 7 days. The active dose is 0.72 mg four times daily for Days 1-5, for a total daily dose of 2.88 mg. Doses on Days 6 and 7 will be 1.44 (2 active, 2 placebo capsules) and 0.72 mg (1 active, 3 placebo capsules), respectively.
  Other Names: Lucemyra
  Arms: Lofexidine/Sham Bridge Device
Drug: Placebo — Inactive study drug, encapsulated to look like the active study drug. Participants will receive capsules 4 times daily for 7 days.
  Arms: Active Bridge Device/ Placebo Study Drug; Sham Bridge Device /Placebo Study Drug
Device: Sham Bridge Device — Inactive Bridge Device which is applied and looks identical to the active Bridge Device
  Other Names: Sham NSS-2 Bridge Device
  Arms: Lofexidine/Sham Bridge Device; Sham Bridge Device /Placebo Study Drug

SUMMARY:
The Bridge Device (BD) is a neuromodulator medical device that has been cleared by the FDA for Opioid Use Disorder (OUD) treatment. Importantly, medical devices reviewed by the FDA are cleared (based on safety) rather than approved (based on efficacy), which means the BD did not need to demonstrate efficacy before it became commercially available. As a result, the device was not required to have a sham-controlled trial for FDA clearance and there is no active research, to the investigators' knowledge, that specifically addresses the degree to which opioid withdrawal can be treated through neuromodulation. To rigorously evaluate the efficacy of the BD for treating OUD, the investigators will enroll persons with active OUD, not currently receiving medications for OUD. Participants will be recruited and admitted to the Clinical Research Unit (CRU) for a 2-3 week period. During participants' residential stay, participants will be stabilized for 7-11 days on four times daily morphine (30 mg, SC) and undergo a precipitated withdrawal challenge using the opioid antagonist naloxone, approximately >= 4 days of morphine maintenance. This is a standard practice for the investigators' study and allows the investigators to objectively assess dependence. The BD and study medication will begin following morphine stabilization. Participants will be randomly assigned to one of three conditions (1) active BD with placebo (BD/P), (2) sham BD with lofexidine (SBD/L), or (3) sham BD and placebo (SBD/P). Participants will use the BD for 5 days and will receive study drug for 7 days. Participants will be monitored for an additional 4 days after device removal to determine whether withdrawal resumes. Participants will undergo a second naloxone challenge after removal of the device/capsule completion to verify lack of opioid tolerance and will be encouraged to begin treatment with oral naltrexone followed by extended release naltrexone. Throughout the residential stay, all participants will be given referral to and assisted with engaging in outpatient treatment following study discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Meets Diagnostic and Statistical Manual-5 criteria for Opioid Use Disorder (OUD) (moderate or severe) based upon Mini-International Neuropsychiatric Interview (MINI)
* Provides a urine sample that tests positive for opioids during screening or have evidence of opioid withdrawal
* Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
* No significant psychiatric illnesses besides OUD
* Seeking treatment to stop using illicit opioids
* Willing to comply with the study protocol
* Have no clinically significant chronic medical or surgical disorders or conditions that are judged by the investigators to prevent participation

Exclusion Criteria:

* Pregnant or breast feeding
* Receiving opioid agonist treatment
* Significant medical illness (e.g., insulin dependent diabetes)
* Significant psychiatric illness (e.g., schizophrenia)
* Use of medical cannabis
* Contraindications for use of the Bridge Device, morphine, lofexidine or naloxone (e.g., hemophilia, psoriasis and other skin conditions, a cardiac pacemaker)
* Have evidence of physical dependence on alcohol or benzodiazepines that requires medical detoxification
* Hypotension (diastolic blood pressure of less than 60 mm Hg or systolic blood pressure of less than 90 mm Hg on screening examination)
* Prolonged corrected QT interval interval on screening ECG (defined as >0.44 seconds for males and >0.46 seconds for females)
* Hepatic or renal impairment, as indicated by the following lab results at the screening session:

  * Aspartate aminotransferase or alanine transaminase >3x upper limit of normal (ULN)
  * Total Bilirubin >2x ULN.
  * Creatinine >1.5x ULN.
* Treatment with a strong 2D6 inhibitor (e.g., paroxetine, thioridazine, cinacalcet, bupropion, methotrimeprazine, fluoxetine, midostaurin, propafenone, glycerol phenylbutyrate, halofantrine, cisapride, dacomitinib, orphenadrine, quinidine)
* Have a known allergy to any of the study medications
* Have circumstances that would interfere with study participation (e.g., impending jail)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants retained | Up to 5 days
  The proportion of participants who are retained (dichotomous: retained, not retained) during the 5 day intervention. Greater retention is indicative of a better treatment outcome.
Withdrawal Severity as measured by Clinical Opiate Withdrawal Scale (COWS) peak score | At the end of day 5
  Peak COWS Score (range: 0-48). Lower peak COWS scores are indicative of better withdrawal suppression.
Withdrawal Severity as measured by area under the curve COWS score | At the end of day 5
  Area under the curve COWS scores (range: 0-240). Smaller area under the curve COWS scores are indicative of better withdrawal suppression.
Withdrawal Severity as measured by COWS peak daily score | Up to 5 days
  Peak daily COWS score (range: 0-48). Lower peak daily COWS scores are indicative of better withdrawal suppression.

SECONDARY OUTCOMES:
Proportion of participants retained | At the end of day 9
  The proportion of participants who are retained (dichotomous: retained, not retained) during the 9 day intervention. Greater retention is indicative of better intervention outcome.
Withdrawal severity as measured by the Subjective Opiate Withdrawal Scale (SOWS) peak score | At the end of day 5
  Peak SOWS Score (range: 0-64). Lower peak SOWS scores are indicative of better withdrawal suppression.
Withdrawal severity as measured by area under the curve SOWS score | At the end of day 5
  Area under the curve SOWS scores (range: 0-320). Smaller area under the curve SOWS scores are indicative of better withdrawal suppression.
Withdrawal severity as measured by the SOWS peak daily score | Up to 5 days
  Peak daily SOWS score (range: 0-64). Lower peak daily SOWS scores are indicative of better withdrawal suppression.
Proportion of Participants who initiate naltrexone at the end of the study | At the end of day 9
  The proportion of participants who initiate naltrexone (dichotomous: yes, no) at the end of day 9. A larger proportion of participants is indicative of better naltrexone initiation success.
Number of concomitant medications used | Up to 5 days
  Number of concomitant medications used per day. A smaller number of concomitant medications used per day is indicative of better treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strain, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No